CLINICAL TRIAL: NCT03367949
Title: Assessment of the Accuracy of Surgical Guide Designed From Dental Model Optical Scan Versus Impression Inversion With Markers Techniques in Computer Guided Implantology. Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdullah Ahmed Elmasry, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SGCBCTELMASRY
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Accuracy of Surgical Guide in Computer Guided Implantology
Keywords: Surgical guide; impression inversion; stereolithographic surgical guides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each patient will be given a code by the researcher (A.A) and the observers will be blind to which group this case belong.
  Patients, evaluators and data analyst will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accuracy of surgical guide from Model optical scan (No Intervention)
- Accuracy of surgical guide from Impression inversion Technique (Active Comparator)
  Interventions: Other: Surgical guide designed from Impression inversion with markers

INTERVENTIONS:
Other: Surgical guide designed from Impression inversion with markers — Rather than using optical scan of the cast , We will use impression inversion technique with VPS impression and adding CBCT Markers on the tray
  Arms: Accuracy of surgical guide from Impression inversion Technique

SUMMARY:
Dental model cast accuracy can be affected by many variables as tray material, impression material and time elapsed before pouring the impression. All these factors would affect the accuracy of the surgical guide

Impression inversion with markers technique avoids the dimension changes that may happen from pouring of the dental model cast. Also it saves time as no need for optical scan of the model cast and for scan appliance even in cases of multiple restoration. Adding markers to impression tray ensures an accurate merge even if the patient has restored dentition that may cause scatter during the CT/CBCT scan.

This study will is for Assessment of the Accuracy of Surgical Guide designed from Dental Model Optical Scan versus Impression Inversion with Markers techniques in Computer Guided Implantology.

ELIGIBILITY:
Inclusion Criteria:

1. Partially Edentulous patients seeking for dental implants
2. Patients with Bucco-lingual bone thickness more than 6 mm allowing flapless implant placement.
3. Medically free patients.

   -

   Exclusion Criteria:

1- Patients with thin ridges. 2- Patients with systemic disease that may affect bone quality. 3- Patients with poor oral hygiene and active periodontal diseases. 4- Anatomical situations requiring regenerative procedure. 5- Completely edentulous patient 6-Patient with limited mouth opening

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of angular deviation of virtual implants and actual implant position according to scanning protocol "optical scan of the model" Versus "impression inversion" using CBCT. | Immediate post operative

SECONDARY OUTCOMES:
Evaluation of linear deviation of virtual implants and actual implant position according to scanning protocol " optical scan of the model" Versus " impression inversion " using CBCT | Immediate post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided